CLINICAL TRIAL: NCT06514079
Title: Role of Topical Steroid Injection With Refractory Benign Esophageal Stricture Endoscopic Dilatation in Children
Acronym: ISIs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammad Daboos (Other)
Responsible Party: Sponsor-Investigator, Mohammad Daboos, Professor at Pediatric Surgery Department, Al-Azhar University., Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00012367-24-06-002
Record Dates: First submitted 2024-07-15; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Pediatric Disorder; Esophageal Diseases; Esophageal Stricture
Keywords: Esophageal stricture; Steroid injection; Esophageal dilatation
MeSH Terms: conditions — Esophageal Diseases; Esophageal Stenosis | interventions — Steroids

STUDY DESIGN:
Intervention Model Description: Pediatric patients aged less than 14 years, with refractory benign esophageal strictures and received a dilatation therapy without triamcinolone injections were included in our study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- refractory benign esophageal strictures patients (Experimental): Pediatric patients aged less than 14 years, with refractory benign esophageal strictures and received a dilatation therapy without triamcinolone injections
  Interventions: Procedure: Esophageal dilatation with steroids injection

INTERVENTIONS:
Procedure: Esophageal dilatation with steroids injection — Under general anesthesia with the patient in the left lateral position. A single-channel endoscope was used. Endoscopic bougie dilatation was performed using Wire-guided Polyvinyl dilator Savary Gilliard/SG. Long-acting steroids triamcinolone acetonide was injected via 25-gauge sclerotherapy catheter. One mL solution of triamcinolone acetonide 40mg/ml was diluted with one mL of saline, in a 2 mL disposable syringe, and 0.5 mL each was injected at the proximal margin of the stricture in four quadrants, 2 mL solution in four quadrants
  Other Names: ISIs Endoscopic dilatation

SUMMARY:
This clinical trial study included 21 children with refractory benign esophageal strictures. Upper GI endoscopy performed up to the area of stricture, esophageal dilatation done, endoscopy repeated, and steroid injected intralesional under direct endoscopic vision. The effect of the procedure was followed over a period of 12 months by evaluation of number of dilatation, maximum dilator size, periodic dilatation index (PDI) and dysphagia score.

DETAILED DESCRIPTION:
Background and study aims: Benign esophageal strictures are primarily treated with dilation therapy, but strictures can recur or can be unresponsive, requiring additional or repeated treatment. This study investigates the efficacy and safety of intralesional steroid injections (ISIs) in addition to dilation in patients with refractory benign esophageal strictures.

Methods: This clinical trial study included 21 children with refractory benign esophageal strictures. Upper GI endoscopy performed up to the area of stricture, esophageal dilatation done, endoscopy repeated, and steroid injected intralesional under direct endoscopic vision. The effect of the procedure was followed over a period of 12 months by evaluation of number of dilatation, maximum dilator size, periodic dilatation index (PDI) and dysphagia score.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged less than 14 years
* with refractory benign esophageal strictures
* received a dilatation therapy without triamcinolone injections

Exclusion Criteria:

* failure to pass a guide wire secondary to pharyngeal stenosis
* tracheo-esophageal fistula
* those who received triamcinolone injections at early dilatation

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Maximum dilatation size | 12 months
  achieving a diameter of 11 mm for patients aged <2 years, 12 mm for patients aged between 2 and 5 years, and 15 mm for children aged >5 years with complete relief of symptoms without requiring endoscopic procedure or surgical intervention for at least 6 months

SECONDARY OUTCOMES:
dysphagia score | 12 months
  Dysphagia was graded into the following:
  * Score 0 - No dysphagia: able to eat a normal diet.
  * Score 1 - Moderate passage: able to eat some solid foods.
  * Score 2 - Poor passage: able to eat only semi-solid foods.
  * Score 3 - Very poor passage: able to swallow only liquids only.
  * Score 4 - No passage: unable to swallow anything

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Daboos, Principal Investigator — Department of pediatric surgery, faculty of medicine , Al-Azhar University
Locations (1):
- Mohammad Daboos, Cairo, Select, Egypt